CLINICAL TRIAL: NCT01610011
Title: Acute Glycine Pharmacodynamic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Marc J. Kaufman, Director, Translational Imaging Laboratory, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2010P001576
Record Dates: First submitted 2012-05-28; First posted 2012-06-01 (Estimated); Results first posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Schizophrenia; Psychotic Disorders; N-methyl-D-aspartate receptor; Glycine augmentation; Glycine; Glycine Pharmacodynamics; Glycine Bioavailability; Magnetic Resonance Spectroscopy; Glycine Decarboxylase; Glycine Decarboxylase Mutation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hyperglycinemia, Nonketotic | interventions — Glycine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glycine administration (Experimental): Glycine will be administered once orally to all subjects to determine brain and plasma pharmacodynamics.
  Interventions: Dietary Supplement: Glycine administration

INTERVENTIONS:
Dietary Supplement: Glycine administration — Glycine will be administered once as a 250 cc lemon-flavored beverage based on each subject's body weight. The drink concentration will be 0.4 g/kg glycine (not to exceed 30 grams). Subjects will have 10 minutes to consume the beverage.
  Other Names: Aminoacetic Acid; Aminoethanoic Acid

SUMMARY:
The purpose of this study is to use proton magnetic resonance spectroscopy (MRS) at 4 Tesla to measure brain glycine levels noninvasively at baseline and for 2 hours after a single oral dose of a concentrated glycine-containing beverage, and to compare MRS glycine measurements to glycine blood levels in samples obtained after each MRS spectrum.

The investigators hypothesize that they will observe a high correlation between the magnitude increases in brain and plasma glycine levels over this time frame.

The investigators also hypothesize that we will observe large intersubject variability in glycine uptake rates into brain and blood.

The investigators also hypothesize that subjects with a glycine decarboxylase (GLDC) mutation (triplication) will have lower baseline plasma and brain glycine levels and will experience smaller brain and plasma glycine increases after glycine consumption than controls or family members without the GLDC mutation.

DETAILED DESCRIPTION:
High doses of glycine (0.4-0.8 g/kg/day) administered orally along with certain antipsychotic medications can improve negative symptoms of schizophrenia (e.g., Heresco-Levy et al., 1999). The therapeutic effect appears to be due to glycine's co-agonist activity at glutamatergic N-methyl-D-aspartate receptors, which may correct the glutamatergic hypofunction associated with schizophrenia (e.g., Bergeron et al., 1998). Unfortunately, the therapeutic benefits of orally administered glycine are variable, in part because gut glycine absorption and resultant plasma (and presumably brain) glycine increases are variable (Silk et al., 1974). Even with intravenous glycine administration, which bypasses variability contributed by gut absorption and metabolism, between-subject variability in cerebrospinal fluid (CSF) glycine increments is large (D'Souza et al., 2000), suggesting that brain glycine uptake, metabolism, and turnover differ substantially among individuals.

If brain glycine increments after oral glycine dosing are highly variable, those manifesting smaller or more transient brain glycine increments may not experience clinically significant effects. As a result, glycine's therapeutic efficacy could be underappreciated. Indeed, a multi-site glycine trial in schizophrenia subjects concluded that glycine is not a "…generally effective therapeutic option for treating negative symptoms or cognitive impairments", but included the caveat that "…it is not known if efficacy would have been achieved at substantially higher serum glycine levels" (Buchanan et al., 2007).

Accordingly, we believe that it is important to fully characterize glycine's brain and plasma pharmacodynamic variability, which we will do in healthy subjects and in several members of a family with some members possessing a mutation in their glycine decarboxylase gene (GLDC), which may be associated with abnormal baseline brain and plasma glycine levels and increments after glycine administration. We will use an MRS method we developed to detect brain glycine increases after high-dose oral glycine administration (Prescot et al., 2006; Kaufman et al., 2009) along with standard analytical methods to determine plasma glycine levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult males
* Members of a family known to the research team with some members possessing a GLDC genetic mutation

Exclusion Criteria:

* Contraindications to magnetic resonance scanning including metallic surgical implants or claustrophobia
* History of head injury with loss of consciousness > 5 minutes
* Brain structural abnormalities identified on MRI scan
* Known sensitivity or allergy to glycine
* History of taking glycine or other dietary supplements
* Healthy controls: history of psychiatric or substance use disorders; individuals taking prescription medications
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc J. Kaufman, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Imaging Center, McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Heresco-Levy U, Javitt DC, Ermilov M, Mordel C, Silipo G, Lichtenstein M. Efficacy of high-dose glycine in the treatment of enduring negative symptoms of schizophrenia. Arch Gen Psychiatry. 1999 Jan;56(1):29-36. doi: 10.1001/archpsyc.56.1.29. PMID 9892253
- [Background] Bergeron R, Meyer TM, Coyle JT, Greene RW. Modulation of N-methyl-D-aspartate receptor function by glycine transport. Proc Natl Acad Sci U S A. 1998 Dec 22;95(26):15730-4. doi: 10.1073/pnas.95.26.15730. PMID 9861038
- [Background] Silk DB, Kumar PJ, Perrett D, Clark ML, Dawson AM. Amino acid and peptide absorption in patients with coeliac disease and dermatitis herpetiformis. Gut. 1974 Jan;15(1):1-8. doi: 10.1136/gut.15.1.1. PMID 4820629
- [Background] D'Souza DC, Gil R, Cassello K, Morrissey K, Abi-Saab D, White J, Sturwold R, Bennett A, Karper LP, Zuzarte E, Charney DS, Krystal JH. IV glycine and oral D-cycloserine effects on plasma and CSF amino acids in healthy humans. Biol Psychiatry. 2000 Mar 1;47(5):450-62. doi: 10.1016/s0006-3223(99)00133-x. PMID 10704956
- [Background] Buchanan RW, Javitt DC, Marder SR, Schooler NR, Gold JM, McMahon RP, Heresco-Levy U, Carpenter WT. The Cognitive and Negative Symptoms in Schizophrenia Trial (CONSIST): the efficacy of glutamatergic agents for negative symptoms and cognitive impairments. Am J Psychiatry. 2007 Oct;164(10):1593-602. doi: 10.1176/appi.ajp.2007.06081358. PMID 17898352
- [Background] Prescot AP, de B Frederick B, Wang L, Brown J, Jensen JE, Kaufman MJ, Renshaw PF. In vivo detection of brain glycine with echo-time-averaged (1)H magnetic resonance spectroscopy at 4.0 T. Magn Reson Med. 2006 Mar;55(3):681-6. doi: 10.1002/mrm.20807. PMID 16453318
- [Background] Kaufman MJ, Prescot AP, Ongur D, Evins AE, Barros TL, Medeiros CL, Covell J, Wang L, Fava M, Renshaw PF. Oral glycine administration increases brain glycine/creatine ratios in men: a proton magnetic resonance spectroscopy study. Psychiatry Res. 2009 Aug 30;173(2):143-9. doi: 10.1016/j.pscychresns.2009.03.004. Epub 2009 Jun 24. PMID 19556112
- See also: Brain and Behavior Research Foundation - Awarding NARSAD Grants — http://bbrfoundation.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Glycine Administration GLDC Mutation Subjects: Glycine will be administered once orally to all subjects to determine brain and plasma pharmacodynamics. Glycine administration: Glycine will be administered once as a 250 cc lemon-flavored beverage based on each subject's body weight. The drink concentration will be 0.4 g/kg glycine (not to exceed 30 grams). Subjects will have 10 minutes to consume the beverage.
Period: Overall Study
Arm/Group | Glycine Administration | Glycine Administration GLDC Mutation Subjects
Started | 19 | 2
Completed | 9 | 2
Not Completed | 10 | 0

BASELINE CHARACTERISTICS:
Population: Subjects eligible to undergo magnetic resonance spectroscopy scans and consume a glycine-enriched beverage, who completed both procedures.
Groups:
- Glycine Administration GLDC Subjects: Glycine will be administered once orally to all subjects to determine brain and plasma pharmacodynamics.
  Glycine administration: Glycine will be administered once as a 250 cc lemon-flavored beverage based on each subject's body weight. The drink concentration will be 0.4 g/kg glycine (not to exceed 30 grams). Subjects will have 10 minutes to consume the beverage.
- Total: Total of all reporting groups
Arm/Group | Glycine Administration | Glycine Administration GLDC Subjects | Total
Number analyzed (Participants) | 9 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (11.5) | 48 (19.8) | 35.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 8 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Brain Glycine Increments After Oral Glycine Administration Measured With MRS as Glycine/Total Creatine, Normalized to the Glycine Dose Administered (g/kg).
Description: Brain and plasma glycine levels are measured with proton magnetic resonance spectroscopy at 4T and analytically, respectively. Because glycine doses were limited to 30 g to avoid nausea and vomiting, some subjects with higher weights were administered lower doses per body weight of glycine (g/kg). Therefore, we corrected MRS data by the actual glycine dose administered (g/kg) to account for dosing differences.
Time Frame: For up to 2 hours
Population: Subjects completing the magnetic resonance spectroscopy study.
Measure: Mean (Standard Error); unit: Percent brain glycine/creatine increase
Units Other Than Participants: Peak dose-normalized glycine increase
Groups:
- Glycine Administration Controls; Glycine Administration GLDC Mutation Subjects: Glycine will be administered once orally to all subjects to determine brain and plasma pharmacodynamics.
  Glycine administration: Glycine will be administered once as a 250 cc lemon-flavored beverage based on each subject's body weight. The drink concentration will be 0.4 g/kg glycine (not to exceed 30 grams). Subjects will have 10 minutes to consume the beverage.
Arm/Group | Glycine Administration Controls | Glycine Administration GLDC Mutation Subjects
Number analyzed (Participants) | 9 | 2
Number analyzed (Peak dose-normalized glycine increase) | 9 | 2
Percent brain glycine/creatine increase | 393 (50) | 677 (117)

ADVERSE EVENTS:
Arm/Group | Glycine Administration Controls | Glycine Administration GLDC Mutation Subjects
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/2
Other Adverse Events (participants affected / at risk) | 0/11 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glycine Administration Controls (N=11) | Glycine Administration GLDC Mutation Subjects (N=2)
Any adverse event (Gastrointestinal disorders) | 0 | 0 — 13 subjects were administered glycine and at risk, 11 who provided usable MRS data to complete the study. The remaining 10 subjects were screened but not administered glycine, and thus were not at risk.

LIMITATIONS AND CAVEATS:
This trial was limited by small sample sizes, especially in the GLDC mutation group, since this is a rare genetic mutation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No